CLINICAL TRIAL: NCT07217717
Title: A Phase 3, Multicenter, Prospective Open-Label Study of the Diagnostic Performance of [¹⁸F]FAPI-74 PET/CT for the Detection of Metastatic Disease in Adults With Pancreatic Ductal Adenocarcinoma
Brief Title: Using 18F-FAPI PET to Detect Metastatic Disease in Patients That Have Pancreatic Ductal Adenocarcinoma (PDAC)
Acronym: FAPI-PRO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SOFIE (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18FFAPI-2025P3-PDAC
Record Dates: First submitted 2025-10-14; First posted 2025-10-16 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-01

CONDITIONS: Pancreatic Ductal Adenocarcinoma (PDAC)
Keywords: PDAC; FAP; FAPI; PET; Fibroblast Activation Protein; Fibroblast Activation Protein Inhibitor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with pancreatic ductal adenocarcinoma receiving [18F]FAPI-74 (Experimental)
  Interventions: Drug: [18F]FAPI-74 PET/CT

INTERVENTIONS:
Drug: [18F]FAPI-74 PET/CT — [18F]FAPI-74 is a radioactive diagnostic agent indicated for use with Positron Emission Tomography (PET) imaging for the detection of Fibroblast Activation Protein (FAP) positive cancer cells and cancer-associated fibroblasts (CAF) in patients with pancreatic ductal adenocarcinoma.

SUMMARY:
This is a multi-site, open-label, non-randomized, single dose study to assess the clinical utility of [¹⁸F]FAPI-74 PET/CT in the detection of metastatic disease in individuals with pathologically confirmed pancreatic ductal adenocarcinoma. Following screening, using a standardized administration protocol and dose, participants will undergo [¹⁸F]FAPI-74 PET/CT screening. SOC procedures and interventions will be captured during 3 months +/-14 days post injection. The primary objective is to evaluate the sensitivity and specificity of such [¹⁸F]FAPI-74 PET/CT using a composite SOT panel. The maximum expected duration of the trial is approximately 24 months from first patient screening to last patient SOC follow up. The participants will be followed-up for safety for 24 to 72 hours after the dose of [¹⁸F]FAPI-74 PET/CT.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults ≥ 18 years.
* Participants with confirmed PDAC, undergoing staging evaluation for treatment planning.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤2:
* Provided signed, written informed consent obtained prior to any study-related procedures.
* Participants are required to have a ceCT scan of chest, abdomen and pelvis as per standard clinical practice and practice guidelines either 21 days or less prior to entry or planned within 21 days of [¹⁸F]FAPI-74 administration.
* For women who are not postmenopausal (two years of amenorrhea) or surgically sterile (absence of ovaries and/or uterus): agreement to use medically accepted, highly effective methods of contraception (e.g., hormonal implants, combined oral contraceptives, vasectomized partner , during the trial intervention period.

Exclusion Criteria:

* Unequivocal evidence of metastases at the time of enrollment that would preclude surgery as a treatment option.
* Known hypersensitivity to [¹⁸F]FAPI-74.
* Administration of another investigational therapeutic or diagnostic product within 30 days prior to [¹⁸F]FAPI-74 administration.
* Prior administration of a radiopharmaceutical within 10 half-lives of that product from the time of [¹⁸F]FAPI-74 administration.
* Previous cancer diagnosis (except basal cell carcinoma of the skin or in situ carcinoma of the cervix/uterus). Participants treated with curative intent and disease-free for more than 5 years are permitted.
* Hepatic function: T. bili >1.5X ULN or alk phos, ALT, or AST >5X ULN
* Renal function: GFR < 30 mL/min
* Pregnant or breast feeding (a negative pregnancy test is required in women of childbearing potential)
* Inability to undergo the PET/CT scanning procedure.
* Inflammatory bowel disease (Crohn's disease or ulcerative colitis)
* Sarcoidosis
* Treatment, including chemotherapy, radiation or surgery for curative intent of PDAC.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity for detection of distant metastatic disease (M1) using a composite SOT as reference | Time Frame: From enrollment to the end of treatment after 3 month follow up
  To evaluate the diagnostic performance of [¹⁸F]FAPI-74 PET/CT scan in determining the presence or absence of metastatic disease (M1) in patients with pancreatic ductal adenocarcinoma compared with a composite standard of truth (SOT).

SECONDARY OUTCOMES:
Incidence and severity of adverse events using CTCAE v5. | 24-72 hours post-injection
  To assess the safety profile of [¹⁸F]FAPI-74 PET/CT.
Cohen's kappa for pairwise evaluation of inter- and intra-reader agreement | From enrollment to the end of treatment after 3 month follow up
  To assess inter-and intra-reader variability in image interpretation of the presence of metastatic disease
Number of participants with treatment-related adverse events as assessed by body temperature changes | 24-72 hours post-injection
  To assess the safety profile of [¹⁸F]FAPI-74 PET/CT.
Number of participants with treatment-related adverse events as assessed by blood pressure changes | 24-72 hours post-injection
  To assess the safety profile of [¹⁸F]FAPI-74
Number of participants with treatment-related adverse events as assessed by respiration rate | 24-72 hours post-injection
  To assess the safety profile of [¹⁸F]FAPI-74
Number of participants with treatment-related adverse events as assessed by pulse rate | 24-72 hours post-injection
  To assess the safety profile of [¹⁸F]FAPI-74

CONTACTS AND LOCATIONS:
Overall Officials: Sherly Mosessian, Ph.D, Study Director — Sofie Co.
Locations (6):
- United States (6):
  - Helios CR Inc./RadNet, Cerritos, California
  - Hoag Memorial Hospital, Irvine, California
  - Indiana University Health University Hospital, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - UMass/Shields, Worcester, Massachusetts
  - Kettering, Kettering, Ohio

IPD SHARING:
Plan to Share IPD: No